CLINICAL TRIAL: NCT00048607
Title: A Double-Blind, Multicenter, Placebo and Active-Controlled, Acute Extension Study of 2 Doses of MK-0869 in the Treatment of Patients With Major Depressive Disorder
Brief Title: Treatment of Patients With Major Depressive Disorder With MK0869 (0869-062)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0869-062; Formally-65MBS4W; MK0869-062; 2006_408
Record Dates: First submitted 2002-11-04; First posted 2002-11-05 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: aprepitant
  Other Names: MK0869
Drug: Comparator: paroxetine HCL
Drug: Comparator: Placebo (Unspecified)

SUMMARY:
A clinical study to determine the efficacy and safety of MK0869 in the treatment of depression

DETAILED DESCRIPTION:
The duration of treatment is 8 weeks.

ELIGIBILITY:
Patients with Major Depressive Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2002-07-30 (Actual); Primary Completion 2003-12-31 (Actual); Study Completion 2003-12-31 (Actual)

PRIMARY OUTCOMES:
HAMD-17 total score at week 8. Tolerability. | at week 8

SECONDARY OUTCOMES:
CGI-I Scale score at week 8 and Sheehan Disability Scale at week 8 | at week 8

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Keller M, Montgomery S, Ball W, Morrison M, Snavely D, Liu G, Hargreaves R, Hietala J, Lines C, Beebe K, Reines S. Lack of efficacy of the substance p (neurokinin1 receptor) antagonist aprepitant in the treatment of major depressive disorder. Biol Psychiatry. 2006 Feb 1;59(3):216-23. doi: 10.1016/j.biopsych.2005.07.013. Epub 2005 Oct 24. PMID 16248986
- [Background] Liu KS, Snavely DB, Ball WA, Lines CR, Reines SA, Potter WZ. Is bigger better for depression trials? J Psychiatr Res. 2008 Jul;42(8):622-30. doi: 10.1016/j.jpsychires.2007.07.003. Epub 2007 Sep 7. PMID 17825841
- Available data/document: CSR Synospis Link — http://www.merck.com/clinical-trials/policies-perspectives.html